CLINICAL TRIAL: NCT01053780
Title: Effects of Remote Intercessory Prayer in Outcomes of Pregnants Women: a Randomized Controlled Trial
Brief Title: Effects of Remote Intercessory Prayer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UNESC
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2009-10

CONDITIONS: Remote Intercessory Prayer
Keywords: Intercessory Prayer, pregnants

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Intercessory Prayer — A committed group of six people selected by the chief investigator prayed nine consecutive days for the patients in the intervention group; they were blind to the identity , the patients' first name, were given to the intercessors.
Behavioral: Intercessory Prayer — A committed group of six people selected by the chief investigator prayed nine consecutive days for the patients in the intervention group; they were blind to the identity , the patients' first name, were given to the intercessors.

SUMMARY:
Intercessory prayer can improve the outcome of pregnancies?

ELIGIBILITY:
Inclusion Criteria:

* be pregnant, belong to the public health system

Exclusion Criteria:

* no consent to participate in the research

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 565 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Apgar score | birth . The time to collect the outcome must be at least the tenth day after making randomization. If the birth occurs before the patient will be excluded from the study.

SECONDARY OUTCOMES:
type of delivery complications in childbirth | birth or abortion. There isn't a pre-determined time. Must be at least 9 days after randomization to allow time to be done the intervention (intercessory prayer)

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Maria Inês da Rosa, Criciúma, Santa Catarina
  - Universidade do Extremo Sul Catarinense, Criciúma, Santa Catarina